CLINICAL TRIAL: NCT05067517
Title: A Double Blind, Randomized, Placebo-controlled Trial Evaluating the Efficacy and Safety of Nintedanib Over 52 Weeks in Patients With Progressive Fibrosing Coal Mine Dust-Induced Interstitial Lung Disease (PF-CMD-ILD)
Brief Title: Efficacy & Safety of Nintedanib in Patients With Progressive Fibrosing Coal Mine Dust-Induced Interstitial Lung Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to enroll any subjects. IRB closed study in agreement with PI.
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012199067
Record Dates: First submitted 2021-07-22; First posted 2021-10-05 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Progressive Fibrosing Interstitial Lung Disease
Keywords: Coal Mine Dust
MeSH Terms: interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nintedanib (Active Comparator): Nintedanib 150 mg administered PO twice daily
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator): Placebo administered PO twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib — Randomized in a 1:1 ratio to either oral nintedanib 150 mg (n=80) or matching placebo (n=80) twice daily.
  Other Names: OFEV
  Arms: Nintedanib
Drug: Placebo — Randomized in a 1:1 ratio to either oral nintedanib 150 mg (n=80) or matching placebo (n=80) twice daily.
  Arms: Placebo

SUMMARY:
Assess efficacy (as measured by annual rate of decline in FVC) and safety. The hypothesis is that nintedanib will be safe and effective therapy for patients with progressive fibrosing CMD-ILD over a period of 52 weeks. Test Article - Nintedanib 150 mg administered PO twice daily or matching placebo. A total of 160 patients meeting inclusion/exclusion criteria will be randomized in a 1:1 ratio to either oral nintedanib 150 mg (n=80) or matching placebo (n=80) twice daily. A randomization scheme will be used that balances the group for potential confounders (proportion with PMF or small opacity-only PF-CMD_ILD and proportion of ever- or never-smokers). The dose of the study drug may be reduced to 100 mg twice daily or interrupted temporarily to manage adverse events (AEs).

DETAILED DESCRIPTION:
This is a single center, prospective, randomized, double-blind, placebo-controlled study to investigate the efficacy and safety of nintedanib in patients with progressive fibrosing CMD-ILD over 52 weeks. The study will be led by and based at the West Virginia University School of Medicine and the West Virginia Clinical and Translational Science Institute (WVCTSI) and will recruit participants regionally, including from its associated Practice-Based Network of 24 healthcare systems and 94 individual clinics. Recruitment will also be sought in collaboration with Dr. Cohen from federally-funded Black Lung Clinics across the region and from partner CTSAs at the University of Kentucky and University of Virginia. It is planned to randomize a total of 160 patients in a 1:1 ratio to either oral nintedanib 150 mg (n=80) or matching placebo (n=80) twice daily. The dose of the study drug may be reduced to 100 mg twice daily with subsequent increase back to full dose or interrupted temporarily to manage adverse events (AEs). For each patient, the study will consist of two parts: part A and part B. The duration of part A, a randomized prospective controlled double-blinded trial, will be 52 weeks.

Following completion of the week 52 visit, patients will continue to have study visits every 16 weeks (Part B) until the last patient completes 52 weeks. In part B, patients will remain on blinded therapy with continued data collection.

In part A, patients will attend screening study visits (-4 to -2 weeks) and then at 0, 4, 8, 12, 24, 36, and 52 weeks. In addition, telehealth visits will be conducted at visits 2, 18, 30, 44, and 51 weeks via phone by the study coordinator. Part B visits will take place at 16 week intervals until study completion (last patient completes 52 weeks). To reduce the amount of missing data, patients who discontinue the trial drug (for any reason) prior to completing the 52-week treatment period will be asked to attend all visits and undergo all examinations as originally planned. In addition, for patients who prematurely discontinue trial medication and are unable to complete the scheduled visits, every attempt will be made to collect information on vital status at week 52 and at the time of data cut-off for the primary data analysis and at the conclusion of part B. It is estimated that patient recruitment will take up to 24 mos.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent consistent with International Conference on Harmonization Tripartite Guideline for Good Clinical Practice (ICH-GCP) and local laws signed prior to entry into the study (and prior to any study procedure including shipment of pre- existing High Resolution Computer Tomography (HRCT), spirometry or other medical records to reviewer).
* Male or female patients aged >= 18 years at Visit 1.
* Progressive Fibrosing Coal Mine Dust-Induced Interstitial Lung Disease (PF-CMD- ILD) based on a history of at least 5 years' work in surface or underground coal mining and presence of Progressive Massive Fibrosis (PMF) within 24 months of screening visit; or small opacity pneumoconiosis plus decline in percent predicted FVC of > 5% relative to high quality spirometry performed 12-24 months prior to screening visit, as assessed by the investigator.
* Pneumoconiotic changes documented on screening chest HRCT. Must include large opacities consistent with PMF or small opacities consistent with pneumoconiosis (as described previously).
* Carbon Monoxide Diffusion Capacity (DLCO) corrected for Hemoglobin (Hb) ≥ 30% and <80% predicted of normal at screening visit.
* FVC >= 45% predicted at screening visit.

Exclusion Criteria:

* For those with PMF and past spirometry data, stable lung function based on a fall in percent predicted FVC of < 5% relative to most recent high quality spirometry obtained at least 12 months but no more than 5 years prior to screening
* Continued employment in a job such as active mining associated with ongoing coal mine dust or respirable crystalline silica dust exposure.
* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) > 1.5 x Upper Limit of Normal (ULN) at screening visit.
* Bilirubin > 1.5 x ULN at screening visit.
* Creatinine clearance <30 mL/min calculated by Cockcroft-Gault formula at screening visit.
* Patients with underlying chronic liver disease (Child Pugh B or C hepatic impairment). Child Pugh A patients may be enrolled and started at a dose of 100mg BID

  * Previous treatment with nintedanib or pirfenidone.
  * Other investigational therapy received within 1 month or 6 half-lives (whichever was greater) prior to screening visit.
* Use of any of the following medications for the treatment of Interstitial Lung Disease (ILD): azathioprine (AZA), cyclosporine, MMF, tacrolimus, oral corticosteroids (OCS) >20mg/day and the combination of OCS+AZA+NAC within 4 weeks of Visit 2, cyclophosphamide within 8 weeks of Visit 2, rituximab within 6 months of screening visit. The eligible patients with comorbid rheumatoid arthritis (RA) or other connective tissue diseases (CTD) is expected to be on disease- modifying anti-rheumatic drug (DMARD) e.g. methotrexate or TNF inhibitors. All approved RA/CTD medications are allowed at stable doses at baseline and during the study.
* Diagnosis of Idiopathic Pulmonary Fibrosis (IPF) based on American Thoracic Society (ATS)/ European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) 2011 Guidelines.
* Significant Pulmonary Arterial Hypertension (PAH) defined by any of the following

  * Previous clinical or echocardiographic evidence of significant right heart failure
  * History of right heart catheterization showing a cardiac index <= 2 l/min/m²
  * PAH requiring parenteral therapy with epoprostenol/treprostinil
* In the opinion of the Investigator, other clinically significant pulmonary abnormalities.
* Major extrapulmonary physiological restriction (e.g. chest wall abnormality, large pleural effusion)
* Cardiovascular diseases, any of the following:

  * Severe hypertension, uncontrolled under treatment (≥160/100 mmHg), within 6 month of Visit 1
  * Myocardial infarction within 6 months of Visit 1
  * Unstable cardiac angina within 6 months of Visit 1
* Bleeding risk, including any of the following:

  * Known genetic predisposition to bleeding.
  * Patients who require

    * Fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, direct thrombin inhibitors, heparin, hirudin)
    * High dose antiplatelet therapy. [Note: Prophylactic low dose heparin or heparin flush as needed for maintenance of an indwelling intravenous device (e.g. enoxaparin 4000 I.U. s.c. per day), as well as prophylactic use of antiplatelet therapy (e.g. acetyl salicylic acid up to 325 mg/day, or clopidogrel at 75 mg/day, or equivalent doses of other antiplatelet therapy) are not prohibited].
  * History of hemorrhagic central nervous system (CNS) event within 12 months of screening visit.
* Any of the following within 3 months of screening visit:

  * Hemoptysis or hematuria
  * Active gastro-intestinal (GI) bleeding or GI - ulcers
  * Major injury or surgery (Investigators judgment).
* Coagulation parameters: International normalized ratio (INR) >2, prolongation of prothrombin time (PT) and activated partial thromboplastin time (aPTT) by >1.5 x ULN at Visit 1.
* History of thrombotic event (including stroke and transient ischemic attack) within 12 months of screening visit.
* Known hypersensitivity to the trial medication or its components (i.e. soya lecithin)
* Patients with peanut allergy.
* Other disease that may interfere with testing procedures or in the judgment of the Investigator may interfere with trial participation or may put the patient at risk when participating in this trial.
* Life expectancy for disease other than ILD < 2.5 years (Investigator assessment).
* Planned major surgical procedures.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Women of childbearing potential not willing or able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly as well as one barrier method for 28 days prior to and 3 months after nintedanib administration. A list of contraception methods meeting these criteria is provided in the patient information. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post- menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy
* In the opinion of the Investigator, active alcohol or drug abuse that will preclude the patient from adhering to the protocol.
* Patients not able to understand or follow trial procedures including completion of self- administered questionnaires without help.
* A study subject may not participate in another research study while participating in this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Annual rate of decline in FVC in mL (absolute) | Baseline after first drug intake (planned post visits with Spirometry test)
  Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Annual rate of decline in FVC in mL (absolute) | 12 weeks after first drug intake (planned post visits with Spirometry test)
  Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Annual rate of decline in FVC in mL (absolute) | 24 weeks after first drug intake (planned post visits with Spirometry test)
  Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Annual rate of decline in FVC in mL (absolute) | 36 weeks after first drug intake (planned post visits with Spirometry test)
  Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Annual rate of decline in FVC in mL (absolute) | 52 weeks after first drug intake (planned post visits with Spirometry test)
  Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible.

SECONDARY OUTCOMES:
FVC change from baseline | 52 weeks after first drug intake (planned post visits with Spirometry test)
  Planned with post visit Spirometry test.
FVC Change from baseline, relative decline % predicted | 52 weeks after first drug intake (planned post visits with Spirometry test)
  Planned with post visit Spirometry test.
Absolute FEV1 annual rate of decline in mL | 52 weeks after first drug intake (planned post visits with Spirometry test)
  Planned with post visit Spirometry test
Relative decline in FEV1 % predicted | 52 weeks after first drug intake (planned post visits with Spirometry test)
  Planned with post visit Spirometry test
Change from baseline in FEV1 change % predicted | 52 weeks after first drug intake (planned post visits with Spirometry test)
  Planned with post visit Spirometry test
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms cough domain score | Baseline
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms cough domain score (cough score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in cough score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline cough score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline cough score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms cough domain score | Week 2
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms cough domain score (cough score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in cough score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline cough score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline cough score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms cough domain score | Week 18
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms cough domain score (cough score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in cough score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline cough score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline cough score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms cough domain score | Week 30
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms cough domain score (cough score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in cough score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline cough score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline cough score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms cough domain score | Week 44
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms cough domain score (cough score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in cough score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline cough score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline cough score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms cough domain score | Week 51
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms cough domain score (cough score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in cough score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline cough score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline cough score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms dyspnea domain score | Baseline
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms dyspnea domain score (dyspnea score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in dyspnea score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline dyspnea score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline dyspnea score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms dyspnea domain score | Week 2
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms dyspnea domain score (dyspnea score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in dyspnea score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline dyspnea score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline dyspnea score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms dyspnea domain score | Week 18
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms dyspnea domain score (dyspnea score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in dyspnea score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline dyspnea score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline dyspnea score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms dyspnea domain score | Week 30
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms dyspnea domain score (dyspnea score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in dyspnea score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline dyspnea score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline dyspnea score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms dyspnea domain score | Week 44
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms dyspnea domain score (dyspnea score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in dyspnea score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline dyspnea score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline dyspnea score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Symptoms dyspnea domain score | Week 51
  Living with Pulmonary Fibrosis (L-PF) questionnaire is a 44 item questionnaire with two modules Symptoms (23 items) and Impacts (21 items) where the symptoms module yields three domain scores dyspnea, cough and fatigue as well as a total symptoms score (impacts module yields a single impacts score). L-PF Symptoms dyspnea domain score (dyspnea score) ranges from 0-100, the higher the score the greater the impairment. If missing items were ≥50 % within a score, then the corresponding score was set to missing. Absolute change from baseline in dyspnea score at week 52 is based on a Mixed Model Repeated Measures, with fixed effects for baseline dyspnea score, HRCT fibrotic pattern, visit, treatment-by-visit interaction, baseline dyspnea score-by-visit interaction and random effect for participant, visit as repeated measure. The Adjusted mean is based on all analyzed participants in the model.
Absolute change from baseline in King's Brief Interstitial Lung Disease Questionnaire (K- BILD) total score | Baseline
  King's Brief Interstitial Lung Disease questionnaire (K-BILD) consists of 15 items and 3 domains: breathlessness and activities, psychological, and chest symptoms. Possible score ranges from 0-100, score of 100 representing the best health status. If missing items were >50% per domain, the domain score was set to missing. If any of the domain scores were missing, the total score was set to missing. Absolute change from baseline in K-BILD Total score at week 52 in the overall population. Mild frustration may be experienced by the participant when completing the questionnaire over the phone with the study coordinator. The participant is allowed to skip questions and not complete the questionnaire if desired.
Absolute change from baseline in King's Brief Interstitial Lung Disease Questionnaire (K- BILD) total score | Week 2
  King's Brief Interstitial Lung Disease questionnaire (K-BILD) consists of 15 items and 3 domains: breathlessness and activities, psychological, and chest symptoms. Possible score ranges from 0-100, score of 100 representing the best health status. If missing items were >50% per domain, the domain score was set to missing. If any of the domain scores were missing, the total score was set to missing. Absolute change from baseline in K-BILD Total score at week 52 in the overall population. Mild frustration may be experienced by the participant when completing the questionnaire over the phone with the study coordinator. The participant is allowed to skip questions and not complete the questionnaire if desired.
Absolute change from baseline in King's Brief Interstitial Lung Disease Questionnaire (K- BILD) total score | Week 18
  King's Brief Interstitial Lung Disease questionnaire (K-BILD) consists of 15 items and 3 domains: breathlessness and activities, psychological, and chest symptoms. Possible score ranges from 0-100, score of 100 representing the best health status. If missing items were >50% per domain, the domain score was set to missing. If any of the domain scores were missing, the total score was set to missing. Absolute change from baseline in K-BILD Total score at week 52 in the overall population. Mild frustration may be experienced by the participant when completing the questionnaire over the phone with the study coordinator. The participant is allowed to skip questions and not complete the questionnaire if desired.
Absolute change from baseline in King's Brief Interstitial Lung Disease Questionnaire (K- BILD) total score | Week 30
  King's Brief Interstitial Lung Disease questionnaire (K-BILD) consists of 15 items and 3 domains: breathlessness and activities, psychological, and chest symptoms. Possible score ranges from 0-100, score of 100 representing the best health status. If missing items were >50% per domain, the domain score was set to missing. If any of the domain scores were missing, the total score was set to missing. Absolute change from baseline in K-BILD Total score at week 52 in the overall population. Mild frustration may be experienced by the participant when completing the questionnaire over the phone with the study coordinator. The participant is allowed to skip questions and not complete the questionnaire if desired.
Absolute change from baseline in King's Brief Interstitial Lung Disease Questionnaire (K- BILD) total score | Week 44
  King's Brief Interstitial Lung Disease questionnaire (K-BILD) consists of 15 items and 3 domains: breathlessness and activities, psychological, and chest symptoms. Possible score ranges from 0-100, score of 100 representing the best health status. If missing items were >50% per domain, the domain score was set to missing. If any of the domain scores were missing, the total score was set to missing. Absolute change from baseline in K-BILD Total score at week 52 in the overall population. Mild frustration may be experienced by the participant when completing the questionnaire over the phone with the study coordinator. The participant is allowed to skip questions and not complete the questionnaire if desired.
Absolute change from baseline in King's Brief Interstitial Lung Disease Questionnaire (K- BILD) total score | Week 51
  King's Brief Interstitial Lung Disease questionnaire (K-BILD) consists of 15 items and 3 domains: breathlessness and activities, psychological, and chest symptoms. Possible score ranges from 0-100, score of 100 representing the best health status. If missing items were >50% per domain, the domain score was set to missing. If any of the domain scores were missing, the total score was set to missing. Absolute change from baseline in K-BILD Total score at week 52 in the overall population. Mild frustration may be experienced by the participant when completing the questionnaire over the phone with the study coordinator. The participant is allowed to skip questions and not complete the questionnaire if desired.
Progression of chest HRCT findings graded according to the International Classification of High-Resolution Computed Tomography for Occupational and Environmental Respiratory Diseases (ICOERD) system | Week 52
  Change in chest HRCT findings graded according to the International Classification of High-Resolution Computed Tomography for Occupational and Environmental Respiratory Diseases (ICOERD) system
6 Minute Walk Test | Week 52
  Change in distance walked from baseline.
Time to all-cause mortality | 52 weeks after first drug intake
  Time to death over 52 weeks defined as the time from date of first drug intake until date of death from any cause for participants with known date of death (from any cause).
Time to respiratory mortality over 52 weeks | 52 weeks after first drug intake
  Time to death due to respiratory cause over 52 weeks is defined as the time from date of first drug intake until date of death attributed to respiratory causes.
Time to progression (defined a ≥10 %absolute decline in Forced Vital Capacity (FVC) % predicted) or death | Over 52 weeks
  Time to progression or death over 52 weeks is defined as the time from date of first drug intake to date of progression, or date of death (from any cause) if a participant died earlier. Date of progression is defined as the date when ≥ 10% of absolute decline in FVC percent predicted compared to baseline occurred for the first time as measured by Spirometry test
Proportion of patients with a relative decline from baseline in FEV1 and/or FVC % predicted of more than 10 percent at week 52 | Up to 52 weeks after first drug intake
  Measured with Spirometry test over the course of study
Proportion of patients with a relative decline from baseline in FEV1 and/or FVC % predicted of more than 5 percent at week 52 | Up to 52 weeks after first drug intake
  Measured with Spirometry test over the course of study
Proportion of patients with an absolute decline from baseline in FVC % predicted of >10% at week 52 | Week 52
  Measured with Spirometry test over the course of study
Proportion of patients with an absolute decline from baseline in FVC % predicted of >5% at week 52 | Week 52
  Measured with Spirometry test over the course of study
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) Total score at week 52 | Week 52
  The cough symptom score will be calculated using the living with pulmonary fibrosis questionnaire (L-PF). L-PF cough symptom score ranges from 0 to 92; the higher the score, the greater the impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Sangani, MD, Principal Investigator — West Virginia University